CLINICAL TRIAL: NCT00771069
Title: A Retrospective, Multi Centre, Non-interventional, Observational Study to Investigate Treatment Pattern of Blood Pressure in the Type II Diabetes Mellitus Patients With DM Related Complication and Hypertension.
Brief Title: Hypertensive Treatment Pattern Survey for Type II Diabetes Mellitus Patients With Complication and Hypertension
Acronym: CRYSTAL-CO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-CKR-DUM-2008/3
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension
Keywords: Hypertension; Type II DM; DM related complication; JNC7; 2007 ESH-ESC guidelines; survey
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Type II Diabetes Mellitus patients with Complication and Hypertension

SUMMARY:
This study will address the treatment rate and control rate of hypertension, treatment pattern and factors to affect blood pressure control by examining (retrospective) medical records of Type II DM patients with DM related complication and hypertension, among outpatients coming to the Endocrinology Department in 20 general hospital settings nationwide.

ELIGIBILITY:
Inclusion Criteria:

* After diagnosed type II DM, patients received treatment for a least 3 years
* Type II DM patients with hypertension and its complication.
* Visited out-patients to care center after 1 Jan. 2008

Exclusion Criteria:

* Secondary hypertension patients
* Patients not receiving hypertension medication
* Patients stopping BP medication, by physician's order
* Patients currently enrolled in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type II Diabetes Mellitus patients with Complication and Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Attainment rate to the target blood pressure. | After collecting all Patient Record Form.

SECONDARY OUTCOMES:
Attainment to the target blood pressure will be investigated according to DM related complications. | After collecting all Patient Record Form.
Change in the DBP/SBP value will be investigated according to the DM Complication | After collecting all Patient Record Form.
Treatment pattern and factors that affect BP control | After collecting all Patient Record Form.

CONTACTS AND LOCATIONS:
Overall Officials: Joonwoo Bahn, Study Director — Astrazenca Korea
Locations (13):
- South Korea (13):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Sungnam, Gyeonggi-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Jeonju, Keollabuk
  - Research Site, Busan
  - Research Site, Deagu
  - Research Site, Deajeon
  - Research Site, Incheon
  - Research Site, Kwangju
  - Research Site, Seoul